CLINICAL TRIAL: NCT06884644
Title: Analysis of Local and Systemic Oxygen Saturation During Monotonous Exercise Using the Example of 'Death by Squats'
Brief Title: Local and Systemic Oxygen Saturation During 'Death by Squats' Exercise
Status: Recruiting | Type: Observational
Sponsor: Bundeswehr University Munich (Other)
Responsible Party: Principal Investigator, Annette Schmidt, PhD, Prof. Dr. Annette Schmidt, Bundeswehr University Munich
Other Study IDs: DBS23
Record Dates: First submitted 2025-02-08; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Oxygen Saturation; Fatigue; Anaerobic Threshold; Quadriceps Muscle
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Death by Airsquat Exercise: All participants follow the exercise protocol, based on the "every minute on the minute" principle:
  Starting off with 10 body weight squats in the first minute (after completion, the remaining seconds can be always be used as a break). In minute two, 12 squats have to be completed. In minute three, 14 squats, and so forth. Until maximum exertion is reached and/or until the number of squats within 60 seconds can not be increased further. Every individual stops at his/her performance limit
  Interventions: Diagnostic Test: Death by Airsquat

INTERVENTIONS:
Diagnostic Test: Death by Airsquat — Increasing number of squats have to be completed every minute (EMOM principle).

SUMMARY:
During the exercise intervention "Death by Squats", which compasses body weight squats until maximum exertion, 25-30 subjects shall be tested for heart rate, the oxygen saturation of the vastus medialis and the triceps, resting and at maximum exertion blood lactate, as well as the rate of perceived exertion on the borg scale. At the end, all should indicate their primary reason for stopping (local fatigue, systemic fatigue, time constraints, motivational deficit).

DETAILED DESCRIPTION:
Subjects in this study will be measured while they are engaged in an exercise protocol until maximum exertion, each in groups of three persons. The overall duration of the study is planned from April 2023 (start of recruitment) until December 2024 (finalization of data acquisition and analysis).

Subjects are executing a CrossFit workout which is planned as follows: Every minute, participants have to perform a given number of Airsquats (bodyweight squat). The first minute starts off with 10 repetitions, the remaining time can be used as a break. In minute two, 12 repetitions have to be done, in minute three 14 repetition, and so on. The subjects stick to this protocol until maximum exertion, in other words, until they are no longer able to execute the given repetitions within the actual minute. During the workout, heart rate is tracked by a 'Polar' chest strap, and the oxygen saturation of the vastus medialis and the triceps are measured using the 'Moxy' muscle oxygen monitor. Further, at rest and at maximum exertion, a blood lactate sample is taken (EKF lactate scout). Subjects rate their perceived exertion on the borg scale after quitting and indicate their primary reason for stopping (local fatigue in legs, systemic fatigue, time constraints).

ELIGIBILITY:
Inclusion Criteria:

* being moderately to severely physically active al least 2 hours/week (all types of sport are eligible)

Exclusion Criteria:

* akute infections, musculoskeletal injuries
* chronic cardiovascular or pulmonary diseases (in case of uncertainty, we recommend appraisal from medical personnel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female participants of 18 years and older, that are performing a CrossFit class with the EMOM workout "Death by Airsquat".
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Local and systemic SmO2 curve | From the start of the exercise intervention until individual exhaustion (expected between 15 to 30 minutes), with SmO₂ continuously recorded during exercise and final measurement taken immediately upon exhaustion.

SECONDARY OUTCOMES:
Type of sports practiced | Questionnaire administered within 5 minutes after test completion to assess type of sports practiced.

OTHER OUTCOMES:
Anthropometric parameters will be assessed | Anthropometric measurements will be taken immediately after the completion of the exercise intervention (expected between 15 to 30 minutes after the start of exercise).
  The following anthropometric parameters will be assessed:
  * body mass (kg)
  * body height (cm)
  * BMI (kg/m², calculated from body mass and height)
  * limb circumference (cm)
  * skinfold thickness (mm)
Blood lactate concentration at rest and post-exercise | At rest (prior to exercise) and immediately upon individual exhaustion (expected between 15 to 30 minutes after the start of exercise). Additional post-exercise measurements at 2, 5, and 10 minutes if applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Bundeswehr Munich, Munich, Bavaria, Germany